CLINICAL TRIAL: NCT04450121
Title: Comparison Between Fekry and Air-Q Intubating Airways as Conduit for Fibreoptic Endotracheal Intubation in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N 54-2018/Ms
Record Dates: First submitted 2020-01-13; First posted 2020-06-29 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Fekry VS the Air-Q Intubating Airways

STUDY DESIGN:
Intervention Model Description: Comparison between the two airways regarding:
  1. Time to Glottic view.
  2. Grade of bronchoscopic view.
  3. Success of intubation from 1st trial.
Who Masked: Participant, Investigator
Masking Description: Randomization will be done using computer generated number and concealed using sequentially numbered, sealed opaque envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA (n =22) (Active Comparator): Patients will be intubated using Air-Q airway
  Interventions: Device: Patients will be intubated using Air-Q airway
- GF (n =22) (Active Comparator): Patients will be intubated using Fekry airway
  Interventions: Device: Patients will be intubated using Air-Q airway

INTERVENTIONS:
Device: Patients will be intubated using Air-Q airway — Both groups:
  Grade 1: Split airway provides an unobstructed path for bronchoscope from mouth to glottis.
  Grade 2: Tongue rests against posterior pharyngeal wall causing partial obstruction to bronchoscope.
  Grade 3: Epiglottis rests against posterior pharyngeal wall causing partial obstruction to bronchoscope.
  Grade 4: Tongue and epiglottis rest against posterior pharyngeal wall, both causing partial obstruction to bronchoscope.
  Grade 5: Tongue rests against posterior pharyngeal wall causing total obstruction to bronchoscope (failure).
  Grade 6: Epiglottis rests against posterior pharyngeal wall causing total obstruction to bronchoscope (failure)

SUMMARY:
The fibreoptic bronchoscope remains one of the most important methods of intubating patients particularly when there is difficulty with intubation.

Facilitating fiberoptic oropharyngeal intubation procedure, specific airways have been devised to push the tongue anteriorly to clear a passage for the fibrescope into the trachea.

Of these airways the Air-Q Intubating Laryngeal Airway (Air-Q) (Cookgas, St. Louis, MO, USA) and Fekry Oral Intubating Airway (Ameco Technology, Cairo, Egypt).

DETAILED DESCRIPTION:
The Air-Q Intubating Laryngeal Airway (Air-Q):

The Air-Q™ Intubating Laryngeal Airway (Air-Q) (Cookgas, St. Louis, MO, USA) is a SAD that was designed primarily to act as a conduit for the passage of a cuffed tracheal tube during tracheal intubation (1), Compared with the LMA, the Air-Q has a shorter silicon airway tube that allows an easy visualization of vocal cords and intubation and removal of the device after tracheal tube insertion. The device has a removable color coded connector, allows intubation through the airway tube. The device is also wider, C-curved and has an integrated bite block which makes it easier to place reinforces the tube and diminishes the need for a separate bite block, with an elevation ramp that facilitates intubation and directs the tube toward the laryngeal inlet. It also has a built-up mask for improved seal. All of these features facilitate the passage of the tracheal tube through the device and into the trachea.

Fekry airway (Oral Intubating Airway; Egyptian Patent 28118):

Several modifications of oropharyngeal airways aiming to allow facilitation of intubation and easy removal of the airway after placement of ETT.

In Fekry airway, modification of the Williams airway facilitates the airway removal after ETT insertion without need to remove the international part of the ETT (this reduce risk of ETT dislodgement during airway removal).

The modification made to the Williams airway is that the roof of the proximal cylindrical tunnel is opened from its upper part to allow one step insertion of the tube. There is no need for removal of the tube connector after tube insertion. It allows passage of the suction catheter and may allow oxygen insufflations through a catheter.

As mastering airway management in difficult cases is an essential job to anesthesiologist, we think it is important to find an easy adjunct to this hard job.

investigators hypothesized that Fekry airway could offer a better conduit to flexible fiberoptic intubation rather than the air-Q device, because it needs less experience in how to use, less intubation time.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years old.
* Of both sexes.
* With American Society of Anaesthesiologists (ASA) physical status class I-ll.
* Scheduled for elective surgery under general anesthesia requiring ETT placement.

Exclusion Criteria:

* Patient refusal.
* Patient that has any documented or suspected difficult airway or neck or upper respiratory tract abnormalities, facial deformities that invalidate Ganzouri airway score.
* Patient that has any active cardiac or chest problem and risk of aspiration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Endoscopy insertion time | Withen 15 seconds from induction og Generel Anesthesia
  Time from introducing the tip of scope through the proximal end of the airway device or mouth until the visualization of carina (multiple attempts will be added to compute this time

SECONDARY OUTCOMES:
ITHIN Intubation time | Withen 15 seconds from induction og Generel Anesthesia
  Timing of complete intubation
Grade of endoscopic view | Withen 15 seconds from induction og Generel Anesthesia
  Endoscopic view grading
Success rate of intubation from 1st trial | Withen 15 seconds from induction og Generel Anesthesia
  1st trial Success
Score of success of endotracheal intubation | Withen 15 seconds from induction og Generel Anesthesia till Study Completion
  Endotracheal intubation Score of success
Number of intubation and device insertion attempts | Withen 15 seconds from induction og Generel Anesthesia
  Attempts Number of intubation and device insertion
Complications | Withen 15 seconds from induction og Generel Anesthesia
  Coughing, laryngospasm, stridor, hoarseness, bronchospasm, arterial desaturation (SpO2<92), aspiration, bleeding or swelling to the lips, tongue, teeth, or blood staining the airway.

CONTACTS AND LOCATIONS:
Overall Officials: Randa Badawi, M.D, Principal Investigator — Cairo University; Maha M Ismail Youssef, M.D, Principal Investigator — Cairo University; Ahmed Moamen Mahmoud, M.Sc, Principal Investigator — Cairo University; Hany M El-Hadi Shoukat, M.D, Principal Investigator — Cairo University; Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Maha Mohamed Ismail Youssef, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Publication